CLINICAL TRIAL: NCT06004557
Title: Validation d'un Outil numérique d'évaluation Multidimensionnelle Pour Les Personnes âgées Dans un Contexte de Consultations gériatriques
Brief Title: Validation of a Digital Multidimensional Assessment Tool for the Elderly in Geriatric Consultations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RIVAGES (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02818-35
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Elderly People in a Consultation Context
Keywords: Tablet; multidimensional assessment; geriatrics; consultation; Validation of a measurement tool

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to validate a digital multidimensional assessment tool for elderly people in geriatric consultations. The aim is to use a digital tablet to rapidly assess several risks (loss of functional independence, risk of falling, risk of malnutrition, risk of depression and risk of burden for the carer) in the context of hospital consultations.

DETAILED DESCRIPTION:
The use of digital tools on tablets to gather information from patients is on the increase. Numerous computerised tools exist for identifying health problems and have been validated in the medical world. However, there are currently no digital tools adapted to the elderly in a consultation context. In this project, the investigators want to carry out a cross-sectional observational study to assess the validity of a multidimensional assessment tool on a tablet, self-administered by patients or carers, and also the appropriateness of using it with these groups.

Objectives Multidimensional assessment tools have the advantage of enabling several issues to be addressed systematically. In this research, the investigators want to assess the validity of a multidimensional assessment tool in digital format in a population of elderly people and carers. To do this, the investigators intend to use scales that already exist and are usually used in paper format: the ADL and IADL for dependency, the Mini MNA for nutrition, the Cornell and GDS-15 for depression, the mini Zarit for estimating the burden on carers and the Cetaf score and short FES-I for the risk of falling. These assessment tools have been adapted to digital format and brought together to form a comprehensive multidimensional assessment tool.

The investigators' first objective was to assess the validity of this set of scales in digital format compared with their original paper versions, but the investigators also want to measure the acceptability of this assessment tool in a geriatric population and among family carers. In addition, the investigators plan to assess the adaptability of this tool and its compatibility in a geriatric consultation setting. Finally, the investigators want to measure doctors' satisfaction with the collection of this information, as a time-saving tool for these professionals.

Methods Eighty patients and eighty carers will be included in this study, recruited from the geriatric consultation service (outpatient geriatrics department) at Charles Foix Hospital. These will be people aged over 65, and family carers if it is not possible to carry out the test on a self-administered basis.

To do this, the investigators are planning a quantitative study to compare the scores obtained by the digital version of the test with the data described by the doctors in the reports, and in particular the same scales systematically filled in by the medical profession. In addition, the investigators want to analyse what users say and assess their experience of practical issues (grip, legibility, impression of confidentiality when filling in the form in the waiting room, etc.).

Outlook A multi-theme self-questionnaire assessment of elderly people and their carers waiting for a consultation would save professionals time (in terms of completion time and calculation of results), make data more secure, save paper and provide a complete and systematic scan of a number of potentially serious risks.

ELIGIBILITY:
Inclusion Criteria:

* People aged over 65 attending a geriatric consultation (if patient)
* Person agreeing to take part in the study and having signed the letter of consent (if patient)
* Person caring for an elderly person (if family caregiver)
* Someone who visits their relative at least once a week (if family caregiver)
* Person agreeing to take part in the study and to complete the evaluation tool in paper format and on a tablet for their relative (if family caregiver)

Exclusion Criteria:

* Incapacity to consent (if patient)
* Refusal to take part in the study (if patient)
* Person under legal protection (if patient)
* People in palliative care (if patient)
* Person who usually has little contact with the patient (if family caregiver)
* Refusal to take part in the study (if family caregiver)
* Incapacity to consent (if family caregiver)
* Person under legal protection (if family caregiver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We would like to offer this study to patients who come to us with memory problems, in accordance with the inclusion criteria set out above. If they are unable to take part, and if family carers are available, they will be able to fill in the questionnaire on a tablet.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Tests used to compare results between the digital version (tablet) and results from healthcare profession | about 3 months
  Calculation of the interclass correlation coefficient (ICC), a statistical method for estimating the equivalence of scores obtained from electronic versions.
Method used to compare and visualise discrepancies between the results of the digital version (tablet) and the results of healthcare professionals | about 3 months
  Bland and Altman concordance method, graph showing the differences between the scores obtained by the two scales for each observation.

SECONDARY OUTCOMES:
Qualitative assessment | about 3 months
  Final questionnaire to evaluate user experimentation

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires Pitié Salpêtrière - Charles Foix et Sorbonne Université, Ivry-sur-Seine, France